CLINICAL TRIAL: NCT04832438
Title: Phase 2 Study of 9-ING-41, a Glycogen Synthase Kinase 3 Beta (GSK 3β) Inhibitor, Plus Carboplatin in Patients With Advanced, Metastatic Salivary Gland Carcinoma
Brief Title: 9-ING-41 Plus Carboplatin in Patients With Advanced, Metastatic Salivary Gland Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by NCT05010629
Sponsor: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2102
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-09

CONDITIONS: Salivary Gland Carcinoma; Adenoid Cystic Carcinoma; Salivary Gland Cancer; Salivary Gland Neoplasms
Keywords: advanced; metastatic; 9-ING-41; carboplatin; refractory
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic; Neoplasm Metastasis | interventions — 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 9-ING-41 plus carboplatin (Experimental): Patients will receive 9-ING-41 (15 mg/kg IV on Day 1 and Day 4) in addition to carboplatin (AUC 5 IV on Day 1) each of a 21-day cycle
  Interventions: Drug: 9-ING-41; Drug: Carboplatin

INTERVENTIONS:
Drug: 9-ING-41 — 15 mg/kg as intravenous infusion on Days 1 and Day 4 of a 21-day cycle
Drug: Carboplatin — Carboplatin AUC 5 intravenously on Day 1 of a 21-day cycle

SUMMARY:
9-ING-41 is a small molecule potent selective GSK-3β inhibitor with antitumor activity. This study investigates 9-ING-41 in combination with carboplatin chemotherapy in patients with incurable, recurrent or metastatic salivary gland carcinomas (SGC). Patients with advanced SGC (including all histologic subtypes and adenoid cystic carcinoma [ACC]) will receive 9-ING-41 intravenously (IV) along with carboplatin IV at standard dosing together on Day 1, and 9-ING-41 alone on Day 4 of a 21-day cycle. Participants will be enrolled to two histologic cohorts: Cohort 1 will be comprised of those with ACC, and Cohort 2 will include patients with non-ACC SGC (or all other salivary gland cancer histologies). Treatment will continue until progression of disease, death, or discontinuation of therapy for any reason.

DETAILED DESCRIPTION:
9-ING-41 is a small molecule potent selective GSK-3β inhibitor with antitumor activity. It acts through downregulation of NF-κB and decreases the expression NF-κB target genes cyclin D1, Bcl-2, anti-apoptotic protein (XIAP) and B-cell lymphoma-extra large (Bcl-XL) leading to inhibition of tumor growth in multiple solid tumor cell and lymphoma lines and patient derived xenograft (PDX) models. 9-ING-41 may also function as an immune modulatory agent by decreasing checkpoint expression and enhancement of T-cell / NK-cell effector function. This is a phase 2, open-label, non-randomized, single institution study investigating the novel glycogen synthase kinase-3 beta (GSK-3β) inhibitor 9-ING-41 in combination with carboplatin chemotherapy in patients with incurable, recurrent or metastatic salivary gland carcinomas (SGC). The safety of this combination has been established in the Actuate 1801 study. Thirty-one evaluable patients with advanced SGC (including all histologic subtypes and adenoid cystic carcinoma [ACC]) will receive 9-ING-41 intravenously (IV) along with carboplatin IV at standard dosing together on Day 1, and 9-ING-41 alone on Day 4 of a 21-day cycle. Participants will be enrolled to two histologic cohorts: Cohort 1 will be comprised of those with ACC, and Cohort 2 will include patients with non-ACC SGC (or all other salivary gland cancer histologies). Treatment will continue until progression of disease, death, or discontinuation of therapy for any reason.

The primary aim of the study is to assess the overall response rate (ORR) as defined by RECIST v1.1 in the overall study population (including both Cohorts 1 and 2). Secondary aims include assessing progression-free survival (PFS), overall survival (OS), determining safety and tolerability, measuring patient-reported quality of life metrics, and correlating efficacy with molecular and immunologic predictors of response. We hypothesize that the novel combination of a GSK-3β inhibitor with carboplatin chemotherapy will result in an ORR of 25% or greater in this patient population where no approved therapies have been established.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed salivary gland carcinoma (any histologic subtype, including ACC) with evidence of recurrent, metastatic or advanced, unresectable disease.
2. Willing to provide tumor tissue from a diagnostic biopsy or prior surgery.
3. Age 18 years or older
4. ECOG performance status 0-2 (see Appendix A)
5. Participant must have organ and marrow function as defined below within 14 days prior to study registration:

   * leukocytes ≥ 3,000/mcL
   * absolute neutrophil count ≥ 500/mcL
   * hemoglobin ≥ 8.5 g/dL
   * platelets ≥ 75,000/mcL
   * total bilirubin ≤ 2.0 g/dL
   * AST(SGOT)/ALT(SGPT) ≤ 2.5× institutional upper limit of normal
   * creatinine within normal institutional limits OR
   * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
6. Participants must have documentation of a new or progressive lesion on a radiologic imaging study performed within 12 months prior to study registration (progression of disease over any interval is allowed) and/or new or worsening disease-related symptoms within 12 months prior to study registration.
7. Participants must have at least one RECIST v1.1 measurable non-CNS based lesion.
8. Prior systemic therapy: At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (3 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 5.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia or neuropathy). Any number of prior therapies for recurrent/metastatic SGC are permitted (including prior carboplatin exposure).
9. Ability to understand and the willingness to sign a written informed consent document.
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study treatment.
11. Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 90 days after the last dose of investigational product.

Exclusion Criteria:

1. Metastatic disease impinging on the spinal cord or threatening spinal cord compression. Patients that have had previous treatment of disease with impinging on the cord with either surgery or radiotherapy with clinical or radiographic evidence of response or stability are eligible.
2. Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment), and have no evidence of new or enlarging brain metastases.
3. Concurrent administration of other cancer specific therapy or investigational agents during the course of this study is not allowed.
4. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
5. Pregnant or lactating women.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include: basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low-risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease in the last 2 years is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2030-12-18 (Estimated); Primary Completion 2033-06-18 (Estimated); Study Completion 2034-06-18 (Estimated)

PRIMARY OUTCOMES:
Number of evaluable patients with objective response as measured by RECIST version 1.1 | 3-24 months
  Response and progression will be evaluated in this study using the international Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No